CLINICAL TRIAL: NCT04967755
Title: Taipei Tzu Chi Hospital,The Buddhist Medical Fundation
Brief Title: Jing-Si-Herbal-Tea Accelerates SARS-Cov-2 Load Reduction Among COVID-19 Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yao-Kuang Wu (Other)
Responsible Party: Sponsor-Investigator, Yao-Kuang Wu, Director of division of pulmonary and critical care care medicine, Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation
Organization: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-X-045
Record Dates: First submitted 2021-07-13; First posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Coronavirus
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: one group received ordinal treatment and other group combination Jing-Si-Herbal-Tea and ordinal treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Jing-Si-Herbal-Tea(JSHT) (Experimental): Eligible patients were randomized to receive routine treatment alone based on the Novel Coronavirus Interim Guidelines for Clinical Management of SARS-CoV-2 Infection (Eleventh edition 2021) (control group) or the combination of routine treatment and JSHT (1 drink thrice daily for 7 days) (JSHT group) at the discretion of the attending clinicians.
  Interventions: Drug: Jing-Si-Herbal-Tea

INTERVENTIONS:
Drug: Jing-Si-Herbal-Tea — Eligible patients were randomized to receive routine treatment alone based on the Novel Coronavirus Interim Guidelines for Clinical Management of SARS-CoV-2 Infection (Eleventh edition 2021) (control group) or the combination of routine treatment and JSHT (1 drink thrice daily for 7 days) (JSHT group) at the discretion of the attending clinicians. Routine treatment generally consisted of the supportive treatment such as oxygen therapy, antiviral medications and symptomatic therapies. Adherence to the study medications, clinical outcomes, the use of concomitant medications and adverse events were recorded. The following data were collected at admission: demographics, body mass index, smoking history, comorbidities, CURB-65 Score for pneumonia. Hemogram, laboratory testing, chest X-ray, and nucleic acid assays of SARS-CoV-2 were evaluated at admission and after randomization and on 7th day.
  Other Names: Control

SUMMARY:
Chinese herbal medicine Jing si herbal tea can effectively reduce the expression of SARS CoV2 in the throat of infected patients, provide medical discoveries, formulate effective isolation policies of hospitals and homes, count the virus retention, develop effective medical care and protection of medical personnel, and create a win-win situation.

DETAILED DESCRIPTION:
Background:

COVID-19 is caused by Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV2). Studies have pointed out that the traditional Chinese herbal medicine Yinqiao powder has been analyzed by network pharmacology and it may be through Interleukin-6, Mitogen-Activated Protein Kinase 3, Tumor necrosis factor and Tumor protein p53 pathways treat COVID-19 infection [1]. In addition, the clinical case report pointed out that a 38-year-old woman who currently lives in Wuhan was diagnosed by a Chinese physician and given appropriate Chinese herbal medicine. One week later, the patient's symptoms eased and her lungs CT scan showed that her lungs substantive phenomenon has reduction [2].

Aims of the study:

This study is a prospective observational study with the following three purposes.

First, cooperate with the treatment of the domestic temporary diagnosis and treatment guidelines, observe the expression level of the SARS CoV2 virus of the infected patients, and provide the research and development of effective treatment for the future.

Second, observe the clinical information of infected patients and provide effective and reasonable isolation policies in our country.

Third, observe the changes in the expression of the SARS CoV2 virus of the infected patients, and formulate an effective medical personnel protection plan.

Materials and Methods and Innovations:

This study is a prospective observational study with the following three purposes.

First, in accordance with the domestic temporary treatment guidelines, observe the changes in the human immune system and provide research and development of effective future treatments.

Second, using the existing polymerase chain reaction testing equipment of Taipei Tzu Chi hospital to intensively measure the virus negative (Ct ratio :cycle threshold), to observe whether the compound Chinese herbal medicine Jing si herbal tea can effectively reduce the expression of the SARS CoV2 virus in the infected person. Observe the clinical information of infected patients and provide effective and reasonable isolation policies in our country.

Third, the plan for the protection of medical personnel, to detect the contamination of the personnel in the medical care process, the situation of virus retention, and to plan effective medical personnel protection measures.

Expected outcome:

Chinese herbal medicine Jing si herbal tea can effectively reduce the expression of SARS CoV2 in the throat of infected patients, provide medical discoveries, formulate effective isolation policies of hospitals and homes, count the virus retention, develop effective medical care and protection of medical personnel, and create a win-win situation.

ELIGIBILITY:
Inclusion Criteria:

* COVID infection patient and age over eighteen

Exclusion Criteria:

* severe pneumonia needing mechanical ventilation
* severe systemic diseases (i.e., malignancy, autoimmune diseases, liver or renal diseases)
* women during pregnancy or lactation
* participation in clinical trials within 3 months
* known allergies to the investigational medications
* other conditions judged by the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
viral shedding and the decline of acute inflammation | 3 months
  Reverse transcription-polymerase chain reaction Cycle threshold ratio calculation (numerical value) as rising speed and reducing amplitude of C-Reaction protein (mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Tzuchi hospital, Principal Investigator — Taipei Tzuchi hospital
Locations (1):
- Taipei Tzu chi hospital,The Buddhist medical fundation., Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No